CLINICAL TRIAL: NCT06425653
Title: The Effect of Exercise Program Applied to Patients With Scleroderma on Functional Outcomes: A Randomized Controlled Trial
Brief Title: Exercise With Scleroderma Functional Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Gizem Özbudak, Lecturer, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-9T/25
Record Dates: First submitted 2024-05-10; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Scleroderma, Systemic; Scleroderma, Diffuse; Scleroderma, Limited; Hand Rheumatism; Mouth Movement Impaired
Keywords: exercise; hand and mouth functional outcomes; nursing; scleroderma; quality of life
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Scleroderma, Limited; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: In the control group the standard protocol was applied. The standard protocol included routine care and treatment practices conducted by the same physician at the same institution. In the intervention group in addition to the standard protocol, an exercise program intervention was applied and after the initial interview the "Exercise Program DVD" was provided through mobile phone. All patients were evaluated 4 times: at baseline, at the 4th week (first visit), at the 8th week (second visit) and at the 12th week (final visit) after randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Program (Experimental): In the control group the standard protocol was applied. The standard protocol included routine care and treatment practices conducted by the same physician at the same institution. In the intervention group in addition to the standard protocol, an exercise program intervention was applied and after the initial interview the "Exercise Program DVD" was provided through mobile phone. All patients were evaluated 4 times: at baseline, at the 4th week (first visit), at the 8th week (second visit) and at the 12th week (final visit) after randomization
  Interventions: Other: Exercise Program
- Standart Protocol (No Intervention): The standard protocol included routine care and treatment practices conducted by the same physician at the same institution.

INTERVENTIONS:
Other: Exercise Program — In the intervention group in addition to the standard protocol, an exercise program intervention was applied and after the initial interview the "Exercise Program DVD" was provided through mobile phone. All patients were evaluated 4 times: at baseline, at the 4th week (first visit), at the 8th week (second visit) and at the 12th week (final visit) after randomization
  Arms: Exercise Program

SUMMARY:
The study aims to investigate the effects of an exercise program applied to patients with scleroderma on functional outcomes (hand and mouth functional results and quality of life).

DETAILED DESCRIPTION:
Systemic sclerosis (scleroderma) is a significant, rare autoimmune connective tissue disease characterized by autoantibodies, fibrosis of the skin and internal organs, microvascular injury and vascular damage due to endothelial cell activation (Sepulveda et al., 2019; Rosendahl et al., 2022). The term "scleroderma" is derived from two Greek words "sklero" and "derma" meaning hard skin (Bielacka et al., 2017; Singh et al., 2019).

The global prevalence of scleroderma is estimated to be between 0.3 and 40 per 100,000 population (Alhendi et al., 2020; Benz et al., 2021; Sierakowska et al., 2019). The occurrence of systemic sclerosis in women is three to five times and in some literature up to eight times higher than in men. The disease incidence peaks between the ages of 30 and 65 (Sierakowska et al., 2019; Hughes et al., 2020; Alhendi et al., 2020).

Impairment of hand functions is one of the most significant disabilities in patients with scleroderma and is commonly observed (Gregory et al., 2019; Mugii et al., 2019). The skin of the hand thickens with manifestations including fingertip ulcers, swelling of the fingers, raynaud's phenomenon and subcutaneous calcium deposition (Abreu et al., 2023). Deformities such as loss of flexion in the metacarpophalangeal joints, loss of extension in the proximal and distal interphalangeal joints, loss of abduction, flexion of the thumb and wrist movement can occur, leading to contractures and severe impairment of hand functions (Bongi & Rosso, 2016; Vannajak et al., 2014).

Besides hand function impairment, another significant issue in scleroderma is the fibrotic involvement of the connective tissue of the face and mouth. Patients tend to lose facial expression. Sclerosis of the skin around the lips and mouth area causes a reduction in mouth opening (microstomia) and width (microcheilia) in 43% to 80% of cases (Puzio et al., 2019; Uras et al., 2019).

Rehabilitation strategies which play a crucial role in the management of scleroderma, include psychoeducational interventions, exercise therapy, application of physical methods, assistive devices and orthoses; joint protection and energy conservation approaches, dietary interventions and comprehensive multidisciplinary team care programs (Schouffoer et al., 2011). Among these interventions daily hand exercises are specifically mentioned to improve hand movement and function, and also mouth and facial exercises positively affect mouth opening function (Gregory et al., 2019). Hand rehabilitation enhances hand movement, functionality and strength, as well as participation in daily life activities such as self-care, housework, work and recreational activities, thereby improving quality of life (Bongi & Rosso, 2016). Exercises that stretch the mouth and increase mouth opening are reported to prevent the progression of microstomia and reduce limitations in mouth opening (Puzio et al., 2019; Yuen et al., 2012). Some approaches and techniques involving active exercises for managing microstomia are suggested, indicating success with the performance of mandibular movements (Puzio et al., 2019).

Programs that include hand and oral rehabilitation interventions are needed to prevent hand deformities and oral dysfunctions, ensure positive body perception, provide coping strategies and maintain quality of life (Schouffoer et al., 2011; Vannajak et al., 2014). However, individuals with a rare disease such as scleroderma face many challenges, including lack of knowledge about the disease, difficulties in accurate diagnosis and limited treatment and support options. Professional support services that are usually provided to individuals with more common diseases are not available for scleroderma patients (Delisle et al., 2019).

Scleroderma is a chronic disease that affects multiple systems and can present numerous symptoms and complications, impacting individuals physically, psychologically and socially. Therefore, the care of patients with scleroderma requires an interdisciplinary holistic health approach that encompasses both physical and emotional support. The rarity of scleroderma, the fact that many patients live far from physical therapy and rehabilitation clinics or the necessity of continuous participation in a program necessitates the implementation of nurse-led home programs (Murphy et al., 2018).

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were being aged between 18 to 70 years, having no communication problems, being able to speak Turkish and agreeing to participate in the study.

Exclusion Criteria:

* . The exclusion criteria were not having the ability to regularly perform hand and mouth exercises, having undergone hand surgery in the last six months, having open wounds or contractures on the hand, having hand and mouth functional disorders due to reasons other than scleroderma, having no teeth, having all upper and lower teeth as dentures and being included in a rehabilitation program in the last three months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Demographic and disease characteristics of the participants | After 12 weeks
  Of the patients included in the study, 50.0% (22 patients) were in the intervention group and 50.0% (22 patients) were in the control group. 95.5% of the intervention group were women and 4.5% were men, with the control group also comprising 95.5% women and 4.5% men patients. The mean age of the all patients was 51.70 ± 11.11 years. 63.6% of patients in the intervention group and 59.1% of patients in the control group were diagnosed with diffuse cutaneous scleroderma. The mean duration of scleroderma diagnosis of all the patients was 9.54 ± 6.73 years for the intervention group and 9.4 ± 6.20 years for the control group. The majority in both groups (63.6% in the intervention group / 95.5% in the control group) were nonsmokers. Table 1 compares the demographic and disease characteristics of the groups. Groups were similar with regard to the demographic and disease characteristics.

SECONDARY OUTCOMES:
Hand functional outcomes of the participants | After 12 weeks
  Upon examining the final follow-up hand functional outcomes of the intervention and control group patients, it has been observed that there is a statistically significant difference between the groups in terms of the average total score of the Duruöz Hand Scale for all sub-dimensions including kitchen, dressing, cleaning, workplace and other activities, as well as the overall average total score (p<0.05)

OTHER OUTCOMES:
Oral functional results of the participants | After 12 weeks
  The mouth opening measurements at the final follow-up of the intervention and control group patients included in the study are compared in Table 3. A statistically significant difference was found between the final follow-up mouth opening measurement values of the groups (p<0.05)
Quality of life results of the participants | After 12 weeks
  The final follow-up scores of the World Health Organization Quality of Life (WHOQOL) Scale averages for the patients in the intervention and control groups who participated in the study were compared. When all subdomains of the scale were evaluated, it was determined that there was a statistically significant difference between the final follow-up total score averages for the physical, psychological, social and environmental domains of the patients in both the intervention and control groups (p<0.05)

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Özbudak, PhD, Principal Investigator — Trakya University; Serap Özer, PhD, Study Chair — Ege University; Figen Yargucu Zihni, MD, Study Chair — Ege University
Locations (1):
- Gizem Özbudak, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sierra-Sepulveda A, Esquinca-Gonzalez A, Benavides-Suarez SA, Sordo-Lima DE, Caballero-Islas AE, Cabral-Castaneda AR, Rodriguez-Reyna TS. Systemic Sclerosis Pathogenesis and Emerging Therapies, beyond the Fibroblast. Biomed Res Int. 2019 Jan 23;2019:4569826. doi: 10.1155/2019/4569826. eCollection 2019. PMID 30809542
- [Result] Rosendahl AH, Schonborn K, Krieg T. Pathophysiology of systemic sclerosis (scleroderma). Kaohsiung J Med Sci. 2022 Mar;38(3):187-195. doi: 10.1002/kjm2.12505. Epub 2022 Mar 2. PMID 35234358
- [Result] Kowal-Bielecka O, Fransen J, Avouac J, Becker M, Kulak A, Allanore Y, Distler O, Clements P, Cutolo M, Czirjak L, Damjanov N, Del Galdo F, Denton CP, Distler JHW, Foeldvari I, Figelstone K, Frerix M, Furst DE, Guiducci S, Hunzelmann N, Khanna D, Matucci-Cerinic M, Herrick AL, van den Hoogen F, van Laar JM, Riemekasten G, Silver R, Smith V, Sulli A, Tarner I, Tyndall A, Welling J, Wigley F, Valentini G, Walker UA, Zulian F, Muller-Ladner U; EUSTAR Coauthors. Update of EULAR recommendations for the treatment of systemic sclerosis. Ann Rheum Dis. 2017 Aug;76(8):1327-1339. doi: 10.1136/annrheumdis-2016-209909. Epub 2016 Nov 9. PMID 27941129
- [Result] Singh D, Parihar AK, Patel S, Srivastava S, Diwan P, Singh MR. Scleroderma: An insight into causes, pathogenesis and treatment strategies. Pathophysiology. 2019 Jun;26(2):103-114. doi: 10.1016/j.pathophys.2019.05.003. Epub 2019 May 18. PMID 31130325
- [Result] Alhendi FJ, Werth VP, Sollecito TP, Stoopler ET. Systemic sclerosis: Update for oral health care providers. Spec Care Dentist. 2020 Sep;40(5):418-430. doi: 10.1111/scd.12492. Epub 2020 Jul 6. PMID 33448431
- [Result] Benz K, Baulig C, Knippschild S, Strietzel FP, Hunzelmann N, Jackowski J. Prevalence of Oral and Maxillofacial Disorders in Patients with Systemic Scleroderma-A Systematic Review. Int J Environ Res Public Health. 2021 May 14;18(10):5238. doi: 10.3390/ijerph18105238. PMID 34069099
- [Result] Sierakowska M, Doroszkiewicz H, Sierakowska J, Olesinska M, Grabowska-Jodkowska A, Brzosko M, Leszczynski P, Pawlak-Bus K, Batko B, Wiland P, Majdan M, Bykowska-Sochacka M, Romanowski W, Zon-Giebel A, Jeka S, Ndosi M. Factors associated with quality of life in systemic sclerosis: a cross-sectional study. Qual Life Res. 2019 Dec;28(12):3347-3354. doi: 10.1007/s11136-019-02284-9. Epub 2019 Sep 3. PMID 31482431
- [Result] Hughes M, Pauling JD, Armstrong-James L, Denton CP, Galdas P, Flurey C. Gender-related differences in systemic sclerosis. Autoimmun Rev. 2020 Apr;19(4):102494. doi: 10.1016/j.autrev.2020.102494. Epub 2020 Feb 13. PMID 32062031
- [Result] Gregory WJ, Wilkinson J, Herrick AL. A randomised controlled trial of wax baths as an additive therapy to hand exercises in patients with systemic sclerosis. Physiotherapy. 2019 Sep;105(3):370-377. doi: 10.1016/j.physio.2018.08.008. Epub 2018 Sep 5. PMID 30318128
- [Result] Mugii N, Matsushita T, Oohata S, Okita H, Yahata T, Someya F, Hasegawa M, Fujimoto M, Takehara K, Hamaguchi Y. Long-term follow-up of finger passive range of motion in Japanese systemic sclerosis patients treated with self-administered stretching. Mod Rheumatol. 2019 May;29(3):484-490. doi: 10.1080/14397595.2018.1466635. Epub 2018 May 15. PMID 29667474
- [Result] Marcatto de Abreu MF, Landim S, Yuamoto FY, Lins C, Magalhaes EP, Etchebehere M. Screening tool development for hand surgery referrals in systemic sclerosis. Clinics (Sao Paulo). 2023 Aug 17;78:100270. doi: 10.1016/j.clinsp.2023.100270. eCollection 2023. PMID 37597472
- [Result] Maddali-Bongi S, Del Rosso A. Systemic sclerosis: rehabilitation as a tool to cope with disability. Clin Exp Rheumatol. 2016 Sep-Oct;34 Suppl 100(5):162-169. Epub 2016 Jul 4. PMID 27384349
- [Result] Vannajak K, Boonprakob Y, Eungpinichpong W, Ungpansattawong S, Nanagara R. The short-term effect of gloving in combination with Traditional Thai Massage, heat, and stretching exercise to improve hand mobility in scleroderma patients. J Ayurveda Integr Med. 2014 Jan;5(1):50-5. doi: 10.4103/0975-9476.128859. PMID 24812476
- [Result] Puzio A, Przywara-Chowaniec B, Postek-Stefanska L, Mrowka-Kata K, Trzaska K. Systemic sclerosis and its oral health implications. Adv Clin Exp Med. 2019 Apr;28(4):547-554. doi: 10.17219/acem/76847. PMID 30079996
- [Result] Uras C, Mastroeni S, Tabolli S, Masini C, Pallotta S, Teofoli P, Rocco G, Mazzanti C, Abeni D. A comparison between two educational methods in the rehabilitation of the microstomia in systemic sclerosis: a randomized controlled trial. Clin Rehabil. 2019 Nov;33(11):1747-1756. doi: 10.1177/0269215519858395. Epub 2019 Jun 19. PMID 31216880
- [Result] Schouffoer AA, Ninaber MK, Beaart-van de Voorde LJ, van der Giesen FJ, de Jong Z, Stolk J, Voskuyl AE, Scherptong RW, van Laar JM, Schuerwegh AJ, Huizinga TW, Vlieland TP. Randomized comparison of a multidisciplinary team care program with usual care in patients with systemic sclerosis. Arthritis Care Res (Hoboken). 2011 Jun;63(6):909-17. doi: 10.1002/acr.20448. PMID 21312348
- [Result] Yuen HK, Marlow NM, Reed SG, Mahoney S, Summerlin LM, Leite R, Slate E, Silver RM. Effect of orofacial exercises on oral aperture in adults with systemic sclerosis. Disabil Rehabil. 2012;34(1):84-9. doi: 10.3109/09638288.2011.587589. Epub 2011 Sep 27. PMID 21951278
- [Result] Delisle VC, Gumuchian ST, El-Baalbaki G, Korner A, Malcarne VL, Pelaez S, Carrier ME, Pepin M, Thombs BD; Scleroderma Support Group Project Advisory Team. Training and support needs of scleroderma support group facilitators: the North American Scleroderma Support Group Facilitators Survey. Disabil Rehabil. 2019 Oct;41(20):2477-2482. doi: 10.1080/09638288.2018.1467970. Epub 2018 Apr 26. PMID 29696997
- [Result] Murphy SL, Barber MW, Homer K, Dodge C, Cutter GR, Khanna D. Occupational Therapy Treatment to Improve Upper Extremity Function in Individuals with Early Systemic Sclerosis: A Pilot Study. Arthritis Care Res (Hoboken). 2018 Nov;70(11):1653-1660. doi: 10.1002/acr.23522. PMID 29381834